CLINICAL TRIAL: NCT04812483
Title: Immunomodulation in Young and Midlife Adults With Newly Diagnosed Primary Immune Thrombocytopenia (ITP): A Randomized Open Label Trial With High-dose Dexamethasone Versus Eltrombopag and High-dose Dexamethasone
Brief Title: Immunomodulation With Eltrombopag in ITP
Acronym: iROM2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Children's Hospital Basel (Other)
Collaborators: Stiftung zur Förderung medizinischer und biologischer Forschung (Unknown); Novartis Pharmaceuticals (Industry); University of Erlangen-Nürnberg, Department of Biology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-00044; ks19Schifferli
Record Dates: First submitted 2021-03-01; First posted 2021-03-23 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Primary Immune Thrombocytopenia (ITP)
Keywords: eltrombopag; thrombopoietin receptor agonist (TPO-RA); ITP in young and midlife adults
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — eltrombopag; Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized study evaluating the immunomodulatory effects of eltrombopag versus standard high-dose (HD) DXM therapy (1:1) in newly diagnosed ITP.
Masking Description: The laboratory team will be kept blinded regarding information about response or non-response of patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Arm (Other): HD-DXM will be administered orally (40 mg) from day 1-4, followed by Arm 1:
  No planed further treatment. = standard therapy (without eltrombopag)
  Interventions: Drug: standard therapy (without eltrombopag): HD-DXM
- Study Arm (Experimental): HD-DXM will be administered orally (40 mg) from day 1-4, followed by Arm 2:
  The subjects in the experimental arm will be treated with eltrombopag:
  Eltrombopag (Revolade®), 50 mg PO, from day 5-140. Tapering over 1 week (week 21) from day 141-148 with 50 mg every second day. Eltrombopag will be administered on a starting dose of 50mg. After the end of treatment a clinical and laboratory observation follow-up period until week 30 follows.
  Interventions: Drug: Eltrombopag (Revolade®); Drug: standard therapy (without eltrombopag): HD-DXM

INTERVENTIONS:
Drug: Eltrombopag (Revolade®) — Eltrombopag is a thrombopoietin receptor agonist (TPO-RA) indicated in patients with ITP refractory to first-line drugs or lasting more than 6 months. Administration of Eltrombopag (Revolade®), 50 mg PO, from day 5-140. Tapering over 1 week from day 141-148 with 50 mg every second day.
  Arms: Study Arm
Drug: standard therapy (without eltrombopag): HD-DXM — standard therapy (without eltrombopag): HD-DXM administered orally (40 mg) from day 1-4

SUMMARY:
The study aims to investigate immunomodulatory effects of eltrombopag combined with dexamethasone in young and midlife adult patients with newly diagnosed primary Immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
The randomized open lable study aims to investigate immunomodulatory effects of eltrombopag combined with dexamethasone in young and midlife adult patients with newly diagnosed primary ITP. Treatment protocol will be HD-DXM (40 mg PO, day 1-4) with or without eltrombopag (25-50 mg PO, day 5-140) on an outpatient basis. Immunological investigations will be performed before start of treatment and then on week 3, 20 (end of therapy) and 30.

1. Intervention phase:

   Medical history and physical examination including assessment of severe bleeding every week until week 4, every second week until week 20. Complete blood count every week until week 10. For the adjustment of the Thrombopoietin receptor agonist (TPO-RA) dose - every second week until week 20. Immunologic panel at the beginning and at week 3 and 20.
2. Follow-up:

Three clinical visits are scheduled in the follow-up including a complete blood count: at week 22, 24 and 30. Immunologic panel will be done at week 30 (end of study).

High-dose dexamethasone (HD-DXM) will be administered orally (40 mg) from day 1-4, followed by Arm 1 or 2 (1:1 randomization).

Arm 1: Standard Arm No planed further treatment. = standard therapy. In case of non-response after 2 courses of HD-DXM (week 4): cross-over to Arm 2: Start Eltrombopag (Revolade®), 50 mg PO until day 140 (details see Arm 2).

In case of relapse: repeat HD-DXM (40 mg day 1-4), up to a maximal of 3 courses. Time between 2 courses should be minimal 14 days. In case of re-relapse after the third course: cross-over to Arm 2: Start Eltrombopag (Revolade®), 50 mg PO until day 140 (details see Arm 2).

Arm 2: Study Arm Eltrombopag (Revolade®), 50 mg per os, from day 5-140. Tapering over 1 week from day 141-148 with 50 mg every second day.

In case of non-response after 4 weeks on eltrombopag: drop out

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* Newly diagnosed primary ITP according to the definition of Rodeghiero et al. and a risk of platelet count of <30x109/l or risk of severe bleeding
* First-line therapy maximum for 1 week prior to enrolment
* Bleeding severity and quality of life are neither an inclusion nor an exclusion criterion.

Exclusion Criteria:

* Patients previously treated for ITP more than 7 days prior to enrolment (e.g. Steroid, intravenous immunoglobulin (IVIG), platelet infusion)
* Patients treated with second-line drugs prior to enrolment
* Life-threatening bleeding (and inability to sign informed consent)
* Secondary ITP
* Positive family history for ITP
* Presence or history of autoimmune disease as judged by the investigator
* Hepatosplenomegaly in the clinical examination
* Relevant hepatic disease as judged by the investigator
* Presence or history of thromboembolic disease
* Patients with splenectomy
* Women who are pregnant or breast feeding
* Intention to become pregnant during the course of the study
* Lack of safe double contraception
* Any vaccination 2 weeks prior start of the study
* Immunsuppressive and antiplatelet drugs
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, incompetence to judge
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Change in percentual T-regulatory cells (Tregs) | before (Tregs/CD4), at week 3 and at the end of the treatment (week 20)
  Assessment of the percentage of Tregs (Tregs/CD4) in the study arm compared to the standard arm. The Tregs will be defined as CD4+CD25+ CD127+ in the fluorescence-activated cell sorting (FACS).

SECONDARY OUTCOMES:
Change in Th1/Th2 balance | at baseline and weeks 3, 20 and 30
  Change in Th1/Th2 balance will be performed by analysis of immunologic profile (immune cell characteristics, messenger ribonucleic acid (mRNA) of immune cells, cytokines, cytokine concentrations)
Clinical response to eltrombopag therapy | trial duration (baseline to week 30)
  Clinical response to eltrombopag therapy (by assessing need of inpatient daycare and use of rescue treatment)
Platelet response to eltrombopag | at baseline and weeks 6, 20 and 30
  Platelet response to eltrombopag: proportion of subjects achieving a platelet count of ≥50x109/l (complete response, response and no response;Response at each assessment is defined as a platelet count of ≥ 50x109/l).

OTHER OUTCOMES:
Number of Adverse Events | trial duration (baseline to week 30)
  Safety of eltrombopag analyzed by documentation of number of Adverse Events
Severe bleeding | trial duration (baseline to week 30)
  Severe bleeding is defined as bleeding requiring hospital admission and/or blood transfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Schifferli, Dr. med., Principal Investigator — University Children's Hospital Basel, UKBB
Locations (6):
- Switzerland (6):
  - Aarau Cantonal Hospital, Division of Hematology, Aarau
  - University Children's Hospital Basel (UKBB), Basel
  - University Hospital Basel, Division of Hematology, Basel
  - University Hospital Bern, Division of Hematology, Bern
  - Liestal Cantonal Hospital, Division of Hematology, Liestal
  - Lucerne Cantonal Hospital, Division of Hematology, Lucerne